CLINICAL TRIAL: NCT07308600
Title: Integrating Plasma Metagenomics and Host Response for Accurate Diagnosis of Infected Pancreatic Necrosis in a Prospective Multicenter Cohort of Acute Necrotizing Pancreatitis
Acronym: PROMOTE
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: The Affiliated Hospital Of Guizhou Medical University (Other); LiuZhou People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025040636
Record Dates: First submitted 2025-12-04; First posted 2025-12-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Acute Necrotizing Pancreatitis; Infected Pancreatic Necrosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- definite IPN group: A positive culture of pancreatic or peripancreatic necrotic tissue obtained from the first drainage procedure or operation, or the presence of gas in the fluid collection on contrast-enhanced CT.
- clinical sterile pancreatic necrosis(SPN) group: Clinically stable during hospitalization with no intervention indicated and the blinded reviewers, after exhaustive chart review, identified no objective evidence of pancreatic infection.
- definite SPN group: The same specimen remained sterile after standard aerobic, anaerobic, and fungal culture.
- suspected IPN group: (i) Infectious manifestations occurred during hospitalization, but such manifestations could be cured with antibiotics alone without the need of any surgical intervention (ii) Infectious manifestations emerged during the disease course, and definitive indications for surgical intervention were identified; nonetheless, surgical intervention was not performed during hospitalization, which was attributed to factors including the patient's demise; (iii) No infectious signs emerged during the disease course, but the patient died of massive hemorrhage or multiple organ failure before any invasive procedure could be performed.

SUMMARY:
This study is being done to find a faster and more accurate way to tell whether the necrosis in patients with acute necrotizing pancreatitis (ANP) has become infected. In the absence of microbiological confirmation, clinicians often have to initiate empirical antibiotic therapy for suspected pancreatic infection-a practice supported by current guidelines but one that may contribute to antimicrobial resistance. In this study, the investigators will combine metagenomic next-generation sequencing (mNGS) which could improve the accuracy of infected pancreatic necrosis (IPN) diagnosis and host transcriptional response analysis which could discriminate infectious and noninfectious inflammatory syndromes. In a prospective, multicentre, cohort study, 200 consecutive patients ≥ 14 years with ANP will be enrolled at four tertiary hospitals from Novemeber 2025 to December 2026. If validated, this single-blood approach could enable early, pathogen-directed therapy, curtail unnecessary antibiotics and expedite surgical timing in ANP.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed acute necrotizing pancreatitis (Revised Atlanta 2012) within 48 h of symptom onset
2. Age ≥14 years
3. Written informed consent

Exclusion Criteria:

1. Invasive interventions including percutaneous catheter drainage (PCD) and surgical necrosectomy have already been performed prior to admission.
2. Confirmed infection outside of pancreas, including pulmonary infection, urinary tract infection.
3. Pregnancy .
4. Acute recurrent pancreatitis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute necrotizing pancreatitis from Xiangya Hospital Central South University, Affiliated Hospital of Guizhou Medical University, Liuzhou People's Hospital, Hunan University of Medicine General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the integrated mNGS and host-transcription model for identification of IPN. | through study completion, an average of 2 months